CLINICAL TRIAL: NCT06372249
Title: A Phase ll Randomized Controlled Trial of Soluble Fiber for Asthma
Brief Title: A Clinical Trial of Soluble Fiber for Asthma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Northern Arizona University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-249; 2U54MD012388-06 (NIH)
Record Dates: First submitted 2024-04-03; First posted 2024-04-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Consumption and the Gut Microbiome Composition in a Pediatric Asthma Cohort (No Intervention): Participants are asked to complete a dietary recall questionnaire (ASA 24) that evaluates dietary intake in the last 24 hours. Participants are also sent home with a stool kit and instructions to collect a fecal sample for microbiome analysis. The purpose of the study is to better understand the pathways that connect diet and asthma.
- A Phase II Randomized Controlled Trial of Soluble Fiber for Asthma (Placebo Comparator): Participants are asked to fill out a dietary recall questionnaire (ASA 24) to determine eligibility in the study. If eligible, a nasal wash and blood sample will be collected at the first visit. Study drug or placebo will be given to participant after their visit in a randomized double-blinded nature. The participant will also fil out an Asthma Control Questionnaire (ACQ) and be sent home with 3 stool kits for analysis. Participant will turn in one sample after first visit, the second in three weeks, and the last one after the second study visit. At this second study visit, procedures from the first study visit will be repeated.
  Interventions: Drug: Inulin

INTERVENTIONS:
Drug: Inulin — Soluble tapioca starch from Ingredion.
  Other Names: Fruitafit CLR
  Arms: A Phase II Randomized Controlled Trial of Soluble Fiber for Asthma

SUMMARY:
Randomized controlled trial of soluble fiber (NOVELOSETM 3490). Participants will complete an ASA 24 dietary recall questionnaire to access their fiber intake. If eligible for the study, participants will be supplemented to their target fiber dosage with either soluble fiber (NOVELOSETM 3490) or placebo. Collection of blood serum, fecal samples, and nasal wash will aid in analyzing the microbes present in one's gut and how fiber and diet may impact it. Thus, allowing researchers to better understand the pathways that may connect diet and asthma and if it is possible to improve asthma by altering one's diet.

DETAILED DESCRIPTION:
A Phase II randomized, controlled, clinical trial analyzing the impact of increasing fiber intake and the gut microbiome for children with asthma. If eligible, (determined by inclusions/exclusion criteria as well as fiber intake assess by ASA 24) participants will be put into a fiber (NOVELOSETM 3490) or placebo (Maltodextrin) group. Each participant will fil out an Asthma Control Questionnaire (ACQ), collect a nasal wash, and have their blood drawn. Their study medication will be available for them to pick up after their first visit, and they will receive counseling from the Pharmacist on how to implement it into their diet. They will also be sent home with three stool sample kits to be mailed to Northern Arizona University for microbiome analysis. The first kit will be sent within 7 days of their first visit. The second kit will be sent within 2-3 weeks of their first visit. The second study visit will occur 4-6 weeks after the first visit. All the procedures will be repeated again including taking the ASA 24 questionnaire. The participant will send their final kit within 7 days of completing their last visit. Total study time is 6 weeks. This study is minimal risk which includes risk of fecal contamination, discomfort from collecting specimens, discomfort with answering some of the survey questions, and the risks associated with receiving a blood draw. Participants are compensated for their time and receive a portion of their dietary results. There may not be a direct benefit to the participant, but by participating in this research they may help people in the future with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 6-17
* Asthma diagnosis within the last 2 years
* Fractional excretion of exhaled nitric oxide (FeNO) > 50 ppb OR a clinical history of environmental allergies as defined by a positive skin prick or positive specific immunoglobulin E (IgE) tests to aeroallergens
* No emergency department visits in the past 1 month
* Ability to consume a liquid drink of fiber or placebo
* Ability to return for a 4-6 week follow-up visit
* No special or unique diet

Exclusion Criteria:

* Cystic fibrosis
* Bronchiectasis
* Change in asthma medicines other than short acting bronchodilators planned over the next 4-6 weeks
* Baseline estimated daily fiber intake less than or equal to 16 grams as determined by the ASA 24
* Sibling of a participant already enrolled in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity. | 6 weeks
  A total of 84 participants is required to find significant difference of 54 units of Richness at 90% power with a small effect size. Alpha diversity is used to measure the abundance that individual microbes can be observed. Statistical analysis is used to generate the significance of stool sample diversity as well as how many participants are needed to see the marker.

SECONDARY OUTCOMES:
Asthma control. | 6 weeks
  Assessed via Asthma Control Questionnaire. Scores can range from 0 to 6. With a higher score indicating poor asthma control.
Gut microbiome composition. | 6 weeks
  Analysis of gut microbiome using quantitative polymerase chain reaction (qPCR) and analysis of variance (ANOVA).
Nasal inflammatory response. | 6 weeks
  Measured via quantitative polymerase chain reaction (qPCR).
Quantification of circulating short chain fatty acids. | 6 weeks
  Obtained from analysis of fecal specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rank, Principal Investigator — Phoenix Children's
Locations (1):
- Phoenix Children's, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT06372249/Prot_SAP_000.pdf